CLINICAL TRIAL: NCT04855474
Title: Estimating Post-exercise Protein Requirements in Male and Female Endurance Athletes
Brief Title: Protein Requirements in Male and Female Endurance Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IAAO-ETFM
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Increased Metabolic Requirement; Healthy

STUDY DESIGN:
Intervention Model Description: Eight men and eight women will be provided three different amino acid intakes on three separate occasions (metabolic trials) over 8 hours following a 20km run. All protein intakes have an amino acid composition modelled off of the profile of egg protein.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Protein (Experimental): 0.2 g/kg/day of protein provided as crystalline amino acid made after egg protein.
  Interventions: Dietary Supplement: Amino Acid Intake
- Moderate Protein (Experimental): 1.2g/kg/day of protein provided as crystalline amino acid made after egg protein.
  Interventions: Dietary Supplement: Amino Acid Intake
- High Protein (Experimental): 2.0 g/kg/day of protein provided as crystalline amino acid made after egg protein.
  Interventions: Dietary Supplement: Amino Acid Intake

INTERVENTIONS:
Dietary Supplement: Amino Acid Intake — Participants will consume hourly (8 hours) isoenergetic, isonitrogenous beverages containing one of the three protein intakes (0.2g/kg/d, 1.2 g/kg/d, 2.0g/kg/d) assigned in a randomized order between the three metabolic trials. Drinks will be enriched with stable isotope [13C]phenylalanine. The use of stable isotope [13C]phenylalanine will allow for the determination of the fate of AA in the body (incorporation into body protein or oxidation) which can be used to determine protein (AA) requirements.

SUMMARY:
Protein is an essential macronutrient for post-exercise recovery through its ability to provide the amino acid building blocks that support increased rates of muscle and whole body protein synthesis.

Despite the growing understanding of the importance of post-exercise protein in endurance athlete populations, the impact of sex and female menstrual cycle phase on protein metabolism is not fully understood. To date, no studies have examined protein requirements in female endurance trained athletes.

The aim of the proposed study is to utilize the well-established IAAO method to determine protein requirements in endurance trained female and male athletes in a "real-world" and at-home setting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy endurance trained runners. Total weekly running distance of greater than 50km/week and perform endurance exercise for more than 5 hours/week.
* Age 18-35 years old
* Eumenorrheic over last 3 months (one cycle no longer than 42 days and no shorter than 20 days).
* Not using hormonal contraceptives (the pill, implants and injections, hormonal intrauterine devices (IUDs), vaginal ring, skin patch).
* Do not have polycystic ovarian syndrome (PCOS) or other conditions effecting ovarian hormone regularity.
* Not pregnant within the past year.
* Must meet the classification of 'superior' aerobic power for their respective age category based on the ACSM criteria; (women age 20-29 years VO2max >50ml/kg/min and women age 30-35 years VO2max >46ml/kg/min) (men age 20-29 years VO2max >56ml/kg/min and men age 30-35 years VO2max >54ml/kg/min).

Exclusion Criteria:

* Inability to meet health and physical activity guidelines according to the CSEP 'Get Active' Questionnaire (Appendix G).
* Inability to adhere to study protocol requirements relating to diet and exercise (i.e. alcohol and caffeine consumption, training/exercise prior to beginning a study testing day).
* Regular use of tobacco and/or other recreational drugs/banned substances (i.e. growth hormone, testosterone, marijuana).
* Self-reported intentional or unintentional weight loss (past 6 months) or plan to lose weight (>5-10kg).
* Amenorrhea (self-reported) in the past 3 months.
* Fewer than 6 menstrual cycles per year.
* Answering yes to any questions asked within the COVID-19 screening questionnaire until 14 days of being symptom free and/or having a negative COVID-19 test

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Phenylalanine excretion | 8 hours
  13CO2 production in umol/kg/h

SECONDARY OUTCOMES:
Phenylalanine Oxidation | 8 hours
  [13C]phenylalanine oxidation in umol/kg/h
Phenylalanine net balance | 8 hours
  Difference between phenylalanine rate of appearance and disappearance

OTHER OUTCOMES:
Urinary 3-methylhistidine | 8 hours
  Concentration of urine 3-methylhistidine
Protein requirement | 8 hours
  Estimated breakpoint of phenylalanine excretion, phenylalanine oxidation, and phenylalanine net balance

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, Ph.D, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data described in the manuscript will be made available upon request pending application and approval.

REFERENCES:
- [Derived] Williamson E, Fung HJW, Adams C, West DWD, Moore DR. Protein Requirements Are Increased in Endurance-Trained Athletes but Similar between Females and Males during Postexercise Recovery. Med Sci Sports Exerc. 2023 Oct 1;55(10):1866-1875. doi: 10.1249/MSS.0000000000003219. Epub 2023 May 19. PMID 37710376